CLINICAL TRIAL: NCT03625141
Title: A Phase II Two Cohort Study Evaluating the Safety and Efficacy of Cobimetinib Plus Atezolizumab in BRAFV600 Wild-type Melanoma With Central Nervous System Metastases and Cobimetinib Plus Atezolizumab and Vemurafenib in BRAFV600 Mutation-positive Melanoma With Central Nervous System Metastases
Brief Title: A Study Evaluating the Safety and Efficacy of Cobimetinib Plus Atezolizumab in BRAFV600 Wild-type Melanoma With Central Nervous System Metastases and Cobimetinib Plus Atezolizumab and Vemurafenib in BRAFV600 Mutation-positive Melanoma With Central Nervous System Metastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MO39136; 2018-000759-41 (EudraCT Number)
Record Dates: First submitted 2018-08-02; First posted 2018-08-10 (Actual); Results first posted 2024-02-08 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Metastatic Melanoma
MeSH Terms: conditions — Melanoma | interventions — cobimetinib; atezolizumab; Vemurafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1- cobimetinib and atezolizumab (Experimental): Participants with BRAFV600 wild-type disease will be administered cobimetinib on Days 1-21 of each 28-day cycle; and atezolizumab on Days 1 and 15 of each treatment cycle.
  Interventions: Drug: Cobimetinib; Drug: Atezolizumab
- Cohort 2 - cobimetinib, atezolizumab and vemurafenib (Experimental): Participants with BRAFV600 mutation-positive disease will be administered cobimetinib, atezolizumab and vemurafenib in 28-day treatment cycles. Treatment includes a 28-day run-in period where participants will receive cobimetinib and vemurafenib only. Upon completion of the 28-day run-in period, atezolizumab will be added to their treatment regimen.
  Interventions: Drug: Cobimetinib; Drug: Atezolizumab; Drug: Vemurafenib

INTERVENTIONS:
Drug: Cobimetinib — 60 mg (three tablets of 20 mg each) orally (PO) once a day (QD) on Days 1-21 of each 28-day cycle.
  Other Names: Cotellic
Drug: Atezolizumab — Atezolizumab will be given at a fixed dose of 840 mg by intravenous (IV) infusion on Days 1 and 15 of each 28-day cycle.
  Only for cohort 2, no dose of atezolizumab will be given during the run-in period (cycle 1).
  Other Names: Tecentriq
Drug: Vemurafenib — Participants will receive vemurafenib 960 mg (four 240 mg tablets) orally (PO) twice daily (BID) on days 1-21 of the run-in period (cycle 1); thereafter, they will receive vemurafenib 720 mg dose (three 240 mg tablets) PO BID on days 22-28 of cycle 1 and on days 1-28 of all subsequent cycles.
  Other Names: Zelboraf
  Arms: Cohort 2 - cobimetinib, atezolizumab and vemurafenib

SUMMARY:
This study will evaluate the efficacy and safety of cobimetinib plus atezolizumab in participants with BRAFV600 wild-type melanoma with central nervous system (CNS) metastases and of cobimetinib plus atezolizumab and vemurafenib in BRAFV600 mutation-positive melanoma patients with CNS metastases.

ELIGIBILITY:
Inclusion Criteria:

Disease-specific inclusion criteria:

* Histologically confirmed melanoma with radiologically confirmed brain metastases
* Documented BRAFV600 mutation status of melanoma tumour tissue using a validated genetic test.
* Measurable brain metastases
* Prior systemic therapy for metastatic melanoma is allowed with exceptions as detailed in the exclusion criteria
* Prior SRT or surgical therapy of ≤ 10 brain metastases is allowed but prior WBRT is not allowed
* Adverse effects of all prior systemic or local treatment must have either returned to baseline or become stable and manageable prior to initiation of study treatment.

General inclusion criteria:

* Age ≥18 years
* Able to comply with the study protocol, in the investigator's judgment
* ECOG Performance Status ≤ 2
* Life expectancy of > 3 months
* Willing and able to complete health and quality of life questionnaires required by the protocol
* Adequate hematologic and end-organ function
* Female patients of childbearing potential and male patients with partners of childbearing potential must agree to always use two effective forms of contraception during the course of this study and for at least six months after completion of study therapy.
* Male patients must agree to refrain from donating sperm for at least six months after the last dose of cobimetinib

Exclusion criteria:

Disease-specific exclusion criteria:

* Ocular melanoma
* Leptomeningeal involvement
* Uncontrolled tumour-related pain
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage more than once every 28 days.
* Prior WBRT treatment for CNS disease
* Increasing corticosteroid dose during the seven days prior to initiation of study treatment or current dexamethasone or equivalent dose of > 8 mg/day
* Prior treatment with a BRAF or MEK inhibitor
* For patients assigned to Cohort 1 only: prior immunotherapy in the metastatic setting is not allowed. Prior immunotherapy is allowed in the adjuvant setting, provided it is completed ≥ 90 days prior to study treatment initiation.

For patients assigned to Cohort 2 only: prior immunotherapy in either the adjuvant or metastatic setting is not allowed.

* Major surgical procedure other than for diagnosis within four weeks prior to initiation of study treatment, or anticipation of need for a major surgical procedure during the course of the study
* Known hypersensitivity to biopharmaceutical agents produced in Chinese hamster ovary cells or to any formulation component of cobimetinib or atezolizumab or, for patients assigned to Cohort 2 only, vemurafenib
* Any anti-cancer therapy, including chemotherapy, hormonal therapy and radiotherapy, within two weeks prior to initiation of study treatment
* Patients assigned to Cohort 2 only: Concomitant treatment with anticonvulsants other than gabapentin, vigabatrin and levetiracetam
* Patients assigned to Cohort 2 only: acetaminophen is prohibited within seven days prior to initiation of study treatment unless the patient has an absolute contraindication to the to the use of non-steroidal anti-inflammatory drugs (NSAIDs) or aspirin
* Active malignancy (other than melanoma) or a prior malignancy within the past three years

General exclusion criteria:

* Known risk factors for ocular toxicity
* History of clinically significant cardiac dysfunction
* Inability to swallow medications
* Malabsorption condition that would alter the absorption of orally administered medications
* Traumatic injury within two weeks prior to initiation of study treatment
* Prior allogeneic stem cell or solid organ transplantation
* Active or history of autoimmune disease or immune deficiency
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g. bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan
* Uncontrolled diabetes or symptomatic hyperglycaemia
* Any Grade ≥ 3 haemorrhage or bleeding event within 28 days of study treatment initiation
* History of stroke, reversible ischemic neurological defect, or transient ischemic attack within six months prior to study treatment initiation
* Positive human immunodeficiency virus (HIV) test at screening
* Hepatitis B virus (HBV) infection (chronic or acute)
* Active hepatitis C virus (HCV) infection
* Active tuberculosis
* History of severe allergic, anaphylactic or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* Severe infection within four weeks prior to initiation of study treatment
* Signs or symptoms of infection within two weeks prior to initiation of study treatment
* Any serious medical condition or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes the patient's safe participation in, and completion of, the study
* Any psychological, familial, sociological, or geographical condition that may hamper compliance with the protocol and follow-up after treatment discontinuation
* Pregnancy, breastfeeding, or intention of becoming pregnant during the study. Women of childbearing potential must have a negative serum pregnancy test result within seven days prior to initiation of study treatment.
* Treatment with therapeutic oral or IV antibiotics within two weeks prior to initiation of study treatment
* Administration of a live, attenuated vaccine within four weeks prior to initiationof study treatment or anticipation of need for such a vaccine during the study
* Treatment with systemic immunostimulatory agents within 28 days or 5 half-lives of the drug, whichever is shorter, prior to study treatment initiation
* Treatment with systemic immunosuppressive medications within two weeks prior to study treatment initiation
* Treatment with investigational drug within 28 days or 5 half-lives of the drug, whichever is longer, prior to initiation of study treatment
* For patients to be assigned to Cohort 2 only: anticipated use of any concomitant medication during or within seven days prior to initiation of study treatment that is known to cause QT prolongation
* Consumption of foods, supplements, or drugs that are strong or moderate CYP3A4 enzyme inducers or inhibitors at least seven days prior to initiation of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-12-13 (Actual); Primary Completion 2021-06-07 (Actual); Study Completion 2023-04-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (22):
- Brazil (3):
  - Instituto Nacional de Cancer - INCa; Oncologia, Rio de Janeiro, Rio de Janeiro
  - Oncosite - Centro de Pesquisa Clinica Em Oncologia Ltda, Ijuí, Rio Grande do Sul
  - Hospital das Clinicas - UFRGS, Porto Alegre, Rio Grande do Sul
- France (3):
  - CHU de Nantes; Cancéro-dermatologie, Nantes
  - Institut Claudius Regaud; Departement Oncologie Medicale, Toulouse
  - Institut Gustave Roussy; Dermatologie, Villejuif
- Universitätsklinikum "Carl Gustav Carus"; Klinik und Poliklinik fur Dermatologie, Dresden, Germany
- Orszagos Onkologiai Intezet; Borgyogyaszati Osztaly, Budapest, Hungary
- Italy (6):
  - IRCCS Istituto Nazionale Tumori Fondazione Pascale; Oncologia Medica B, Napoli, Campania
  - Istituto Dermopatico dell'Immacolata (IDI)-IRCCS; IV Divisione Oncologica e Dermatologia Oncologica, Rome, Lazio
  - IRCCS Istituto Nazionale Per La Ricerca Sul Cancro (IST); Oncologia Medica A, Genoa, Liguria
  - Irccs Istituto Europeo Di Oncologia (IEO); Oncologia Medica, Milan, Lombardy
  - Azienda Ospedaliero - Universitaria Pisana U.O. Oncologia Medica 2 Universitaria ? Polo Oncologico, Pisa, Tuscany
  - IOV - Istituto Oncologico Veneto IRCCS, Padua, Veneto
- Riga East Clinical University Hospital Latvian Oncology Centre, Riga, Latvia
- Spain (6):
  - Onkologikoa - Instituto Oncológico de Donostia, Donostia / San Sebastian, Guipuzcoa
  - Hospital Clínic i Provincial; Servicio de Hematología y Oncología, Barcelona
  - Institut Catala d Oncologia Hospital Duran i Reynals, Barcelona
  - Hospital General Universitario Gregorio Marañon; Servicio de Oncologia, Madrid
  - Hospital Universitario Virgen Macarena; Servicio de Oncologia, Seville
  - Hospital General Universitario de Valencia; Servicio de oncologia, Valencia
- Universitätsspital Zürich; USZ Flughafen / H13-7-609, Zurich, Switzerland

REFERENCES:
- [Derived] Dummer R, Queirolo P, Gerard Duhard P, Hu Y, Wang D, de Azevedo SJ, Robert C, Ascierto PA, Chiarion-Sileni V, Pronzato P, Spagnolo F, Mujika Eizmendi K, Liszkay G, de la Cruz Merino L, Tawbi H. Atezolizumab, vemurafenib, and cobimetinib in patients with melanoma with CNS metastases (TRICOTEL): a multicentre, open-label, single-arm, phase 2 study. Lancet Oncol. 2023 Dec;24(12):e461-e471. doi: 10.1016/S1470-2045(23)00334-0. Epub 2023 Jul 14. PMID 37459873
- [Derived] Dummer R, Queirolo P, Abajo Guijarro AM, Hu Y, Wang D, de Azevedo SJ, Robert C, Ascierto PA, Chiarion-Sileni V, Pronzato P, Spagnolo F, Mujika Eizmendi K, Liszkay G, de la Cruz Merino L, Tawbi H. Atezolizumab, vemurafenib, and cobimetinib in patients with melanoma with CNS metastases (TRICOTEL): a multicentre, open-label, single-arm, phase 2 study. Lancet Oncol. 2022 Sep;23(9):1145-1155. doi: 10.1016/S1470-2045(22)00452-1. Epub 2022 Aug 5. PMID 35940183

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 21 centers in 7 countries.
Pre-assignment Details: A total of 80 participants were enrolled at 21 centers.
Period: Overall Study
Arm/Group | Cohort 1- Cobimetinib and Atezolizumab | Cohort 2 - Cobimetinib, Atezolizumab and Vemurafenib
Started | 15 | 65
Completed | 0 | 0
Not Completed | 15 | 65
Not completed — Adverse Event | 0 | 2
Not completed — Study Terminated By Sponsor | 1 | 13
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Withdrawal Of Consent | 0 | 1
Not completed — Death | 11 | 47
Not completed — Progressive Disease | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1- Cobimetinib and Atezolizumab | Cohort 2 - Cobimetinib, Atezolizumab and Vemurafenib | Total
Number analyzed (Participants) | 15 | 65 | 80
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.9 (12.5) | 54.4 (13.9) | 55.6 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 24 | 33
  Male | 6 | 41 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 9 | 9
  Not Hispanic or Latino | 11 | 50 | 61
  Unknown or Not Reported | 4 | 6 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 61 | 72
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Intracranial Objective Response Rate (ORR)
Description: Intracranial ORR is defined as the percentage of participants with either a complete response (CR) or a partial response (PR) in their intracranial disease based on two consecutive assessments >= 4 weeks apart. Disease status for this endpoint will be determined by an Independent Review Committee (IRC) in accordance with Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) with modified measurability definition for intracranial lesions (>= 0.5 cm by MRI) and allowing up to five intracranial target lesions. CR is defined as disappearance of all lesions. PR is defined as >=30% decrease in tumor burden, in the absence of CR. The primary endpoint is analyzed on the BRAFV600 mutation positive (Cohort 2) only as the Sponsor had discontinued enrolment into Cohort 1. Data for Cohort 1 was not collected nor analyzed for this outcome measure.
Time Frame: Baseline up to cut of date (approximately 2.5 years)
Population: The evaluable population included all enrolled participants who received study medication and had at least two post-baseline intracranial tumour assessments for response evaluation.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 2 - Cobimetinib, Atezolizumab and Vemurafenib
Number analyzed (Participants) | 56
Percentage of participants | 46.4 [32.99 to 60.26]

2. Secondary Outcome: Extracranial ORR
Description: Extracranial ORR, defined as the percentage of participants with either a CR or PR in their extracranial disease based on two consecutive assessments >=4 weeks apart, as determined by the investigator according to RECIST v1.1.
Time Frame: Baseline up to cut of date (approximately 2.5 years)
Population: The safety population included all participants who received at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1- Cobimetinib and Atezolizumab | Cohort 2 - Cobimetinib, Atezolizumab and Vemurafenib
Number analyzed (Participants) | 15 | 65
Percentage of participants | 20.0 [4.33 to 48.09] | 56.9 [44.04 to 69.15]

3. Secondary Outcome: Overall ORR
Description: Overall ORR, defined as the percentage of participants with either a CR or PR in their overall disease (i.e. including intracranial and extracranial disease) based on two consecutive assessments >= 4 weeks apart, as determined by the investigator according to RECIST v1.1. CR was defined as disappearance of all target and non-target lesions and (if applicable) normalization of tumor marker levels. PR was defined as at least a 30 percent (%) decrease in sum of diameters of all target lesions, taking as reference the baseline sum of diameters, in the absence of CR.
Time Frame: Baseline up to cut of date (approximately 2.5 years)
Population: The safety population included all participants who received at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1- Cobimetinib and Atezolizumab | Cohort 2 - Cobimetinib, Atezolizumab and Vemurafenib
Number analyzed (Participants) | 15 | 65
Percentage of participants | 26.7 [7.79 to 55.10] | 52.3 [39.54 to 64.85]

4. Secondary Outcome: Progression-Free Survival (PFS)
Description: Intracranial, extracranial and overall PFS defined as the time from study treatment initiation to the first occurrence of disease progression or death from any cause, whichever occurs first, as determined by the investigator according to RECIST v1.1.
Time Frame: Baseline up to cut of date (approximately 2.5 years)
Population: The safety population included all participants who received at least one dose of study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1- Cobimetinib and Atezolizumab | Cohort 2 - Cobimetinib, Atezolizumab and Vemurafenib
Number analyzed (Participants) | 15 | 65
Months
  Intracranial | 2.17 [1.74 to 7.98] | 5.78 [5.36 to 7.43]
  Extracranial | 4.21 [1.84 to 12.65] | 10.68 [7.85 to 13.67]
  Overall | 1.81 [1.71 to 3.71] | 5.49 [5.13 to 7.43]

5. Secondary Outcome: Duration of Response (DOR)
Description: Intracranial, extracranial and overall DOR, defined as the time from the first occurrence of a documented objective response based on two consecutive assessments ≥ 4 weeks apart to disease progression or death from any cause (whichever occurs first), as determined by the investigator according to RECIST v1.1. This endpoint is analyzed on the BRAFV600 mutation positive (Cohort 2) only as the Sponsor had discontinued enrolment into Cohort 1. Data for Cohort 1 was not collected nor analyzed for this outcome measure.
Time Frame: Baseline up to cut of date (approximately 2.5 years)
Population: The safety population included all participants who received at least one dose of study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 2 - Cobimetinib, Atezolizumab and Vemurafenib
Number analyzed (Participants) | 65
Months
  Intracranial: number analyzed (Participants) | 32
  Intracranial | 6.7 [5.6 to 9.5]
  Extracranial: number analyzed (Participants) | 37
  Extracranial | 11.6 [9.2 to 13.0]
  Overall: number analyzed (Participants) | 34
  Overall | 7.4 [5.5 to 9.5]

6. Secondary Outcome: Disease Control Rate (DCR)
Description: Intracranial, extracranial and overall DCR, defined as the percentage of participants with a CR or PR or stable disease (SD) at 16 weeks from study treatment initiation, as determined by the investigator according to RECIST v1.1. CR was defined as disappearance of all target and non-target lesions and (if applicable) normalization of tumor marker levels. PR was defined as at least a 30 percent (%) decrease in sum of diameters of all target lesions, taking as reference the baseline sum of diameters, in the absence of CR. SD is defined as neither sufficient shrinkage to qualify for CR or PR nor sufficient increase to qualify for disease progression. Disease progression is defined as >=20% increase in tumor burden. This endpoint is analyzed on the BRAFV600 mutation positive (Cohort 2) only as the Sponsor had discontinued enrolment into Cohort 1. Data for Cohort 1 was not collected nor analyzed for this outcome measure.
Time Frame: At 16 weeks
Population: The safety population included all participants who received at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 2 - Cobimetinib, Atezolizumab and Vemurafenib
Number analyzed (Participants) | 65
Percentage of participants
  Intracranial | 50.8 [38.07 to 63.40]
  Extracranial | 50.8 [38.07 to 63.40]
  Overall | 50.8 [38.07 to 63.40]

7. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from study treatment initiation to death from any cause.
Time Frame: Baseline up to 4 years, 4 months
Population: The safety population included all participants who received at least one dose of study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 2 - Cobimetinib, Atezolizumab and Vemurafenib
Number analyzed (Participants) | 65
Months | 13.40 [10.68 to 16.92]

8. Secondary Outcome: Time to Cognitive Symptom Deterioration
Description: Time from study treatment initiation to cognitive symptom deterioration, defined as a change (>= 10 points on a 0-100 scale) on selected scales of the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-BN20) (visual disorder, motor dysfunction, communication deficit, headaches, seizures and drowsiness).
Time Frame: Up to 48 months
Population: The PRO-evaluable population included all participants who received any amount of any study medication (e.g., atezolizumab, cobimetinib, or vemurafenib) and had a baseline and at least one post baseline PRO assessment in the questionnaire of interest (EORTC QLQ-C30 or EORTC QLQBN20).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1- Cobimetinib and Atezolizumab | Cohort 2 - Cobimetinib, Atezolizumab and Vemurafenib
Number analyzed (Participants) | 13 | 63
Months
  Visual Disorder | 3.75 [1.87 to NA] — Insufficient number of participants with event. | 2.99 [1.41 to 8.74]
  Motor Dysfunction | 1.87 [1.08 to 19.84] | 6.70 [3.94 to 13.90]
  Communication Deficit | 6.44 [2.83 to NA] — Insufficient number of participants with event. | 13.90 [6.54 to 21.13]
  Headaches | NA [1.08 to NA] — Insufficient number of participants with event. | 10.84 [5.55 to NA] — Insufficient number of participants with event.
  Seizures | 8.31 [8.31 to NA] — Insufficient number of participants with event. | NA [17.74 to NA] — Insufficient number of participants with event.
  Drowsiness | 2.83 [1.08 to NA] — Insufficient number of participants with event. | 7.16 [1.94 to NA] — Insufficient number of participants with event.

9. Secondary Outcome: Time to Symptom and Function Deterioration
Description: Time from study treatment initiation to symptom and function deterioration defined as a change (>= 10 points on a 0-100 scale) in fatigue, physical functioning, cognitive functioning, or role functioning as measured by the Fatigue, Physical, Cognitive, Role Functioning scales of the EORTC QLQ-C30.
Time Frame: Up to 48 months
Population: as for outcome 8
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1- Cobimetinib and Atezolizumab | Cohort 2 - Cobimetinib, Atezolizumab and Vemurafenib
Number analyzed (Participants) | 13 | 63
Months
  Physical Functioning | NA [0.99 to NA] — Insufficient number of participants with event. | 11.56 [5.55 to NA] — Insufficient number of participants with event.
  Cognitive Functioning | 11.99 [1.91 to NA] — Insufficient number of participants with event. | 8.25 [5.55 to NA] — Insufficient number of participants with event.
  Role Functioning | 2.83 [1.35 to 6.47] | 4.07 [1.61 to 6.47]
  Fatigue | 1.35 [0.95 to NA] — Insufficient number of participants with event. | 1.45 [1.38 to 6.47]

10. Secondary Outcome: Duration of Stable/Improved Health-related Quality of Life (HRQoL) Scores
Description: Duration of Stable/Improved HRQoL scores as assessed through use of the two-item Global Health Status (GHS)/HRQoL subscale (Questions 29 and 30) of the EORTC QLQ-C30.
Time Frame: Baseline up to cut of date (approximately 2.5 years)
Population: as for outcome 8
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1- Cobimetinib and Atezolizumab | Cohort 2 - Cobimetinib, Atezolizumab and Vemurafenib
Number analyzed (Participants) | 13 | 63
Months | NA [15.21 to NA] — There were an insufficient number of participants with an event. | 6.14 [3.68 to 10.32]

11. Secondary Outcome: Percentage of Participants With Adverse Events
Description: The safety profile of Cobimetinib plus Atezolizumab and Cobimetinib plus Atezolizumab plus Vemurafenib is evaluated in terms of occurrence and severity of AEs. Severity will be determined according to the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 4.0 (NCI CTCAE v4.0)
Time Frame: Baseline up to 4 years, 4 months
Population: The safety population included all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 2 - Cobimetinib and Vemurafenib: There were 5 participants in Cohort 2 administered with cobimetinib and vemurafenib only as they dropped out during the run-in period.
Arm/Group | Cohort 1- Cobimetinib and Atezolizumab | Cohort 2 - Cobimetinib, Atezolizumab and Vemurafenib | Cohort 2 - Cobimetinib and Vemurafenib
Number analyzed (Participants) | 15 | 60 | 5
Participants
  Occurrence | 15 | 60 | 5
  Grade 1 | 1 | 1 | 0
  Grade 2 | 3 | 13 | 1
  Grade 3 | 9 | 35 | 2
  Grade 4 | 1 | 10 | 0
  Grade 5 | 1 | 1 | 2

ADVERSE EVENTS:
Time Frame: Baseline up to 4 years, 4 months
Arm/Group | Cohort 1- Cobimetinib and Atezolizumab | Cohort 2 - Cobimetinib, Atezolizumab and Vemurafenib | Cohort 2 - Cobimetinib and Vemurafenib
All-Cause Mortality (participants affected / at risk) | 11/15 | 47/60 | 3/5
Serious Adverse Events (participants affected / at risk) | 6/15 | 21/60 | 5/5
Other Adverse Events (participants affected / at risk) | 15/15 | 60/60 | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1- Cobimetinib and Atezolizumab (N=15) | Cohort 2 - Cobimetinib, Atezolizumab and Vemurafenib (N=60) | Cohort 2 - Cobimetinib and Vemurafenib (N=5)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Gallbladder rupture (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatitis toxic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Bacterial diarrhoea (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Limbic encephalitis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 1 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash morbilliform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1- Cobimetinib and Atezolizumab (N=15) | Cohort 2 - Cobimetinib, Atezolizumab and Vemurafenib (N=60) | Cohort 2 - Cobimetinib and Vemurafenib (N=5)
Anaemia (Blood and lymphatic system disorders) | 4 (5) | 11 (11) | 1 (1)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 3 (3) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 8 (8) | 0 (0)
Detachment of retinal pigment epithelium (Eye disorders) | 0 (0) | 3 (5) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Keratitis (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 0 (0) | 2 (2) | 1 (1)
Serous retinal detachment (Eye disorders) | 1 (1) | 3 (3) | 0 (0)
Serous retinopathy (Eye disorders) | 0 (0) | 8 (9) | 0 (0)
Uveitis (Eye disorders) | 0 (0) | 3 (4) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 5 (5) | 0 (0)
Visual impairment (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 7 (8) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 5 (6) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 6 (7) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 6 (17) | 29 (60) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 4 (4) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 6 (6) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 14 (22) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 3 (4) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 5 (5) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (4) | 10 (15) | 1 (1)
Asthenia (General disorders) | 4 (5) | 19 (23) | 0 (0)
Chills (General disorders) | 1 (1) | 2 (3) | 0 (0)
Fatigue (General disorders) | 1 (1) | 4 (4) | 0 (0)
Malaise (General disorders) | 1 (1) | 1 (1) | 0 (0)
Mass (General disorders) | 1 (1) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 6 (12) | 0 (0)
Oedema peripheral (General disorders) | 2 (3) | 8 (9) | 0 (0)
Pyrexia (General disorders) | 3 (5) | 26 (56) | 1 (1)
Xerosis (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic cytolysis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 3 (3) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 4 (4) | 0 (0)
Fungal skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Rash pustular (Infections and infestations) | 2 (2) | 2 (3) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 4 (5) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 4 (9) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 13 (26) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 19 (27) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 14 (21) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 11 (13) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 3 (4) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 2 (31) | 28 (78) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 9 (12) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 5 (5) | 0 (0)
Blood magnesium decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 23 (45) | 0 (0)
Thyroxine free increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 4 (5) | 0 (0)
Tri-iodothyronine free decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Cell death (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 5 (5) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 7 (11) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 6 (6) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0)
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 4 (4) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 19 (24) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (6) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 11 (16) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 0 (0)
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 6 (6) | 0 (0)
Headache (Nervous system disorders) | 2 (6) | 8 (13) | 0 (0)
Sciatica (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 3 (3) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 5 (6) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 3 (3) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (6) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (5) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 4 (9) | 18 (21) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (5) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (5) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 11 (16) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 9 (9) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 20 (29) | 0 (0)
Rash follicular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 17 (20) | 1 (1)
Scab (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Vitiligo (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 10 (12) | 0 (0)
Lymphoedema (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Contrast media allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 3 (3) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 3 (3) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 3 (4) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The Sponsor decided to discontinue enrollment into Cohort 1, which was communicated in a Dear Investigator Letter dated 9 July 2019.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2022-03-04): https://cdn.clinicaltrials.gov/large-docs/41/NCT03625141/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-02): https://cdn.clinicaltrials.gov/large-docs/41/NCT03625141/SAP_001.pdf